CLINICAL TRIAL: NCT04954170
Title: Internal Rotation Resistance Test at Abduction and External Rotation: a New Clinical Test for Diagnosing Subscapularis Lesions
Brief Title: Internal Rotation Resistance Test at Abduction and External Rotation
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2013125
Record Dates: First submitted 2021-07-05; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Rotator Cuff Tears
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- RCT patients: Patients suffering from rotator cuff injury
  Interventions: Diagnostic Test: IRRTM; Diagnostic Test: the lift-off test; Diagnostic Test: the belly-press test; Diagnostic Test: the IRLS test; Diagnostic Test: the bear-hug test; Diagnostic Test: IRRT 0°; Diagnostic Test: Diagnostic arthroscopy

INTERVENTIONS:
Diagnostic Test: IRRTM — IRRT at maximal 90° abduction and maximal external rotation is performed with the shoulder at maximal 90° rotation and the elbow flexed to 90° (Fig. 2). The patient is then asked to resist the external rotation force applied perpendicular to the forearm by the investigator. The test is considered positive if the patient could not hold the position or if he or she showed weakness of resisted internal rotation compared with the other side. It should be noted the maximal 90° abduction and maximal external rotation is active range of motion. Passive motion may affect the result of the test because of severe pain.
Diagnostic Test: the lift-off test — The lift-off test is performed by placing the hand of the affected arm on the back (at the position of the midlumbar spine) and asking the patient to internally rotate the arm to lift the hand off the back [9]. The test is considered positive if the patient is unable to lift the arm posteriorly off the back or if he or she performs the lifting manoeuvre by extending the elbow or the shoulder. Weakness is also as a positive result.
Diagnostic Test: the belly-press test — The belly-press test is performed with the arm at the side and the elbow flexed to 90°, by having the patient press the palm into his or her abdomen by internally rotating the shoulder [3, 5]. The test is considered positive (1) if the patient shows a weakness in comparison with the opposite shoulder or (2) the patient pushes the hand against the belly by wrist flexion, despite instruction to the contrary.
Diagnostic Test: the IRLS test — IRLS test is evaluated with the affected arm of the patient was held by the examiner at maximum internal rotation [10]. The back of the hand is then passively lifted away from the body until almost full internal rotation is reached. Then, the patient is asked to actively maintain this position. The test is considered positive when the patient fails to maintain the position and the hand lagged.
Diagnostic Test: the bear-hug test — The bear-hug test is performed with the palm of one side placed on the opposite shoulder and fingers extended and the elbow positioned anterior to the body [3]. The patient is then asked to hold that position when the examiner tried to pull the patient's hand from the shoulder with an external rotation force applied perpendicular to the forearm. The test is considered positive if the patient could not hold the hand against the shoulder or if he or she showed weakness compared with the other side.
Diagnostic Test: IRRT 0° — IRRT at 0° abduction and 0° external rotation is performed with the arm at the side and the elbow flexed to 90° (Fig. 1). The patient is then asked to resist the external rotation force applied by the investigator. The test is considered positive if the patient could not hold the position at the side or if he or she showed weakness of resisted internal rotation compared with the other side. The test is negative if patients only complain of pain.
Diagnostic Test: Diagnostic arthroscopy — At the time of surgery, general anaesthesia was administered and the patient was placed in beach-chair position. A complete arthroscopic exploration of the glenohumeral joint and the subacromial space was performed through a standard posterior portal. The senior author performed a complete arthroscopic exploration. Arthroscopic evaluation of the rotator cuff was considered the gold standard for making the definitive diagnosis. Evaluation of the SSC was carried out with both a 30° arthroscope and a 70° arthroscope.

SUMMARY:
A new clinical test for evaluating subscapularis (SSC) integrity was described, and its diagnostic value was compared with the present SSC tests (the lift-off, bellypress, IRLS and bear-hug tests). The new test is called internal rotation resistance test at abduction and external rotation (IRRT). The test is performed at maximal 90° of abduction and maximal external rotation. Two hundred and thirty-five consecutive patients suffering from rotator cuff injury were evaluated preoperatively. Six tests were performed to assess the function of the SSC: the lift-off, belly-press, IRLS, the bear-hug, IRRT at 0° abduction and 0° external rotation (IRRT0°) and IRRT at maximal 90° abduction and maximal external rotation (IRRTM). Arthroscopic findings were the reference for diagnosing of SSC lesions.

DETAILED DESCRIPTION:
The subscapularis (SSC) provides 50 % of total rotator cuff strength and constitutes the anterior part of force couples of the glenohumeral joint. The advances in shoulder arthroscopy have resulted in improved detection and treatment of subscapularis tendon pathology. The prevalence is between 27 and 30 % in all shoulder arthroscopies and between 49 and 59 % in arthroscopic rotator cuff surgery .

It would be advantageous for the surgeon to be able to diagnose a SSC tear clinically before surgery is performed for rotator cuff tear. Magnetic resonance imaging (MRI) scans of the shoulder have been widely used as a diagnostic tool for predicting the rotator cuff injuries. But preoperative MRI scans do not reliably predict SSC tears, whether conventional MRI or MR arthrography is used. Many clinical tests have been published to evaluate the integrity of SSC. The first of these was the lift-off test by Gerber that was reported to be very reliable in patients with complete SSC tears. The internal rotation lag sign (IRLS) published by Hertel et al. was specific but more sensitive than the lift-off test for assessing the SSC. The belly-press test described by Gerber et al. was modified by other authors who called it the Napoleon sign or the modified belly-press test. Positive belly-press tests were found with upper-third SSC tears. More recently, the bear-hug test was published by Barth et al. and represented the most sensitive test compared with lift-off, belly-press and Napoleon tests. However, Yoon et al. found belly-press test was more sensitive compared with bear-hug test in the most recent study. In our institute, we also performed internal rotation resistance test (IRRT) at 0° abduction and 0° external rotation (IRRT0°, Fig. 1) and IRRT at maximal 90° abduction and maximal external rotation (IRRTM) to investigate the function of SSC. These tests use resisted internal rotation as the shoulder is at different abduction and external rotation degrees.

Although many of these tests are performed, SSC lesions are still underdiagnosed before operation. Because these 6 tests mentioned above have a distinct position and manner, the individual test might imply different severity of SSC lesions. The SSC is stretched out and more extension in the abduction and external rotation position compared with internal rotation position. The purpose of this study is to describe the new clinical test (IRRTM) for evaluating SSC integrity and to compare its diagnostic value with the present SSC tests (the lift-off, belly-press, IRLS and bear-hug tests). The hypothesis was that the IRRTM would be the most sensitive test for detecting tears of the SSC.

ELIGIBILITY:
Inclusion Criteria:

* patients suffering from rotator cuff injury

Exclusion Criteria:

* patients with shoulder stiffness, instability, calcifying tendinitis, previous surgery and on the contralateral shoulder with diseases.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Two hundred and thirty-five consecutive patients including 107 men and 128 women with the mean age 51 ± 18.3 years (range from 26 to 76 years) were evaluated. There were 173 right and 62 left shoulders.
Sampling Method: Non-Probability Sample
Enrollment: 235 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2013-05-31 (Actual); Study Completion 2013-05-31 (Actual)

PRIMARY OUTCOMES:
patient-reported pain | immediately after the test
  patients feeling severe pain when accomplishing the test

CONTACTS AND LOCATIONS:
Overall Officials: Guoqing Cui, Study Chair — Peking University Third Hospital
Locations (1):
- PekingUTH, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No